CLINICAL TRIAL: NCT05659355
Title: Effects of Constraints Induced Movement Therapy Versus Mirror Therapy on Hand Dexterity and Grip Strength in Children With Hemiplegic Cerebral Palsy
Brief Title: Effects of Constraints Induced Movement Therapy Versus Mirror Therapy in Children With Hemiplegic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0730
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Cerebral Palsy; Hemiplegic Cerebral Palsy
Keywords: cerebral palsy; constraints induced movement therapy; mirror therapy
MeSH Terms: conditions — Cerebral Palsy | interventions — Constraint Induced Movement Therapy; Mirror Movement Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Constraint Induced Movement Therapy
  Interventions: Other: Constraint Induced Movement Therapy (CIMT)
- Control Group (Experimental): Mirror Therapy
  Interventions: Other: Mirror Therapy (MT)

INTERVENTIONS:
Other: Constraint Induced Movement Therapy (CIMT) — I will apply CIMT on effected hand to observe the hand dexterity and grip strength
  Other Names: CIMT
  Arms: Treatment Group
Other: Mirror Therapy (MT) — I will apply Mirror Therapy on effected hand to obeserve the hand dexterity and grip strength
  Arms: Control Group

SUMMARY:
The aim of this study is to find Effects of constraints induced movement therapy (CIMT) versus mirror therapy (MT) on hand dexterity and grip strength in children with hemiplegic cerebral palsy.

DETAILED DESCRIPTION:
Although quite number of research has been done on effects of CIMT and mirror therapy but most of the studies included stroke population. There was no literature on comparative effect of both CIMT and Mirror therapy in children with hemiplegic cerebral palsy. This study will be covering specifically cerebral palsy children to have better treatment techniques to be introduced in therapeutic programs of hemiplegic cerebral palsy children.

ELIGIBILITY:
Inclusion Criteria:

* Children of age range 9-14 year
* Children with diagnosed hemiplegic cerebral palsy
* Children who can perform active extension of affected wrist and more than
* two fingers at an angle of more than 10 degrees
* Active abduction of affected thumb at an angle of 10 degrees
* Children who can respond to simple communication-

Exclusion Criteria:

* Children with uncontrolled seizures
* Botulinum toxin injections or orthopedic surgery in the upper or lower
* extremities within the previous 12 months or planned within the study period
* Children with depression who were unable to cooperate in treatment
* Children who are unable to perform active task training

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
9 Hole pegboard test: | 3 months
  The 9 hole peg test is a standardized quantitative assessment used to measure finger dexterity in patients with various neurological diagnosis.
Haptic (Tactile) Recognition Test: | 3 months
  it's a quantitative measure of haptic (tactile) object recognition design to test one's ability to recognize everyday objects across seven sensory attributes using 14 sets of objects. Haptic recognition of everyday objects is quite fast and highly accurate with 96% correctly named: 68% in less than 3 s and 94% within 5 sec.
Hand Dynamometer: | 3 months
  Hand Dynamometer: Hand dynamometer is an evaluation tool that is used to measure isometric grip force. . Once the grip position is adjusted, the user holds the handle and squeezes the handle

CONTACTS AND LOCATIONS:
Overall Officials: Shabana Ashraf, Principal Investigator — Riphah International University
Locations (1):
- Mobility Quest, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No